CLINICAL TRIAL: NCT03620344
Title: The Effect of Bibliotherapy on Parent and Child Knowledge of ADHD and Treatment Follow-up
Brief Title: ADHD/Me Bibliotherapy Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty getting parents to complete follow-up assessments
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2017-4815
Record Dates: First submitted 2018-07-20; First posted 2018-08-08 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADH-Me Book (Experimental): Families in both conditions will be told that they are receiving additional reading materials to help them and their child better understand the ADHD condition and the available options for treating ADHD. Families in both groups will receive the "Understanding ADHD: Information for Parents About ADHD" brochure. Families assigned to this condition will also receive the ADH-Me! book. Written by a pediatrician and health literacy expert, ADH-Me! is an accessible, rhyming narrative that describes an empathetic journey from the perspective of a child learning to live and succeed with ADHD. The book is intended to help families know what to expect from diagnosis through all stages of treatment, while attempting to foster love and support.
  Interventions: Other: ADH-Me Book and ADHD Informational Brochure
- No ADH-Me Book (Sham Comparator): Families in both conditions will be told that they are receiving additional reading materials to help them and their child better understand the ADHD condition and the available options for treating ADHD. Families in both groups will receive the "Understanding ADHD: Information for Parents About ADHD" brochure.
  Interventions: Other: ADHD Informational Brochure Only

INTERVENTIONS:
Other: ADH-Me Book and ADHD Informational Brochure — "Understanding ADHD" information brochure published by American Academy of Pediatrics and a children's book about ADHD condition
  Arms: ADH-Me Book
Other: ADHD Informational Brochure Only — "Understanding ADHD" information brochure published by American Academy of Pediatrics
  Arms: No ADH-Me Book

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD) is one of the most common neurodevelopmental disorders of childhood. It affects approximately 8% of school aged children and is characterized by persistent symptoms of inattention and/or hyperactivity/impulsivity. Typical ADHD assessments primarily involve interviewing the parents and gathering rating scales from parents and teachers. Feedback regarding diagnosis, clinical conceptualization, and treatment recommendations is usually provided by the clinical staff to the child's parents in the absence of the child. Hence, the ADHD diagnosis and repercussions of that diagnosis are often left unexplained to the child. Research has shown that bibliotherapy is an effective educational tool that can be used to help parents discuss ADHD diagnosis and treatment with their child. The aim of this study is to conduct a randomized trial in which tools for parents who are getting their elementary-aged (7 to 10-year-old) children evaluated for ADHD are explored. The evaluations (N=60) will be conducted at the Center for ADHD at Cincinnati Children's Hospital Medical Center (CCHMC) in Cincinnati, OH. Half of the families (n=30) will be randomly assigned to the intervention group, where they will be provided with the child-focused "ADH-Me!" book during the feedback session, and the remaining half will not receive it. All participants will receive a booklet with general information about ADHD and a list of recommendations from the clinicians. Approximately 3 months after their feedback sessions, follow-up surveys will be conducted via telephone to question the parents and children about their ADHD knowledge, as well as about whether they had followed up on the clinicians' recommendations. It is hypothesized that providing families with the ADH-Me! book will increase families' knowledge about ADHD and facilitate the family following up on treatment recommendations.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Meet ADHD criteria based on ADHD evaluation

Exclusion Criteria:

-

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
ADHD Knowledge and Opinion Survey - Revised | 3 months after ADHD evaluation feedback session
  The knowledge portion of the AKOS-R, which consists of 15 true/false items, was modified by the research team for the 7 to 10-year-old children that will participate in this study. The overall readability of the survey was reduced from a 6th grade to a 4th grade level.

SECONDARY OUTCOMES:
Decision-Making Involvement Scale - Parent Report | 3 months after ADHD evaluation feedback session
  The DMIS is a 30-item measure completed by parents that was developed to assess the degree to which children and adolescents (ages 8 to 19 years) are involved in decisions having to do with their chronic illness management.
Decision-Making Involvement Scale - Youth Report | 3 months after ADHD evaluation feedback session
  The DMIS is a 30-item measure completed by children that was developed to assess the degree to which children and adolescents (ages 8 to 19 years) are involved in decisions having to do with their chronic illness management.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for ADHD, Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share.